CLINICAL TRIAL: NCT01733901
Title: Safety and Effectiveness Study of Percutaneous Catheter-based Renal Sympathetic Denervation as a Method of Secondary Prevention for Patients After Percutaneous Coronary Intervention.
Brief Title: Renal Sympathetic Denervation as Secondary Prevention for Patients After Percutaneous Coronary Intervention.
Acronym: RSD4CHD2PRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Qijun Shan, Professor，Director, Cardiac Arrhythmia Group, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21012-SR-132
Record Dates: First submitted 2012-11-09; First posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease; PCI; Renal sympathetic denervation; Hypertension; Diabetes
MeSH Terms: conditions — Coronary Disease; Hypertension; Diabetes Mellitus | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RSD+PCI+Medicine (Active Comparator): We will recruit 300 randomised CHD patients who meet the inclusion criteria. First undergo percutaneous coronary intervention, and then perform the renal artery angiography procedure to confirm anatomy. If renal artery meet the inclusion criteria, give the renal sympathetic denervation. After renal sympathetic denervation traditional secondary prevention of coronary heart disease is recommend. Finally we will conduct a clinic follow-up every six month and a telephone follow-up every three month(Total 24 months).
  Interventions: Procedure: RSD; Procedure: PCI
- PCI+Medicine (Placebo Comparator): We aslo will recruit 300 randomised CHD patients who meet the inclusion criteria. There are no significant differences in age, gender, race, past medical history,personal history and so on between the two groups. In this group we will perform percutaneous coronary intervention firstly, then give traditional secondary prevention of coronary heart disease just like the RSD+PCI+Medicine group. Third we will conduct a clinic follow-up every six month and a telephone follow-up every three month(Total 24 months).
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: RSD — Contrast renal angiography was performed to localize and assess the renal arteries for accessibility and appropriateness for RSD. Once the anatomy was deemed acceptable, the internally irrigated radiofrequency ablation catheter(Celcius Thermocool,Biosense Webster, Diamond Bar, California) was introduced into each renal artery. then was maneuvered within the renal artery to allow energy delivery in a circumferential, longitudinally staggered manner to minimize the chance of renal artery stenosis. About six to nine ablations at 10 W for 1 min each were performed in both renal arteries. During ablation, the catheter system monitored tip temperature and impedance, altering radiofrequency energy delivery in response to a predetermined algorithm.
  Other Names: renal sympathetic denervation; renal denervation; renal ablation
  Arms: RSD+PCI+Medicine
Procedure: PCI — Percutaneous coronary intervention (PCI) is a non-surgical procedure used to treat the stenotic coronary arteries of the heart found in CHD. During PCI, a cardiologist feeds a deflated balloon or other device on a catheter from the inguinal femoral artery or radial artery up through blood vessels until they reach the site of blockage in the heart. X-ray imaging is used to guide the catheter threading. At the blockage, the balloon is inflated to open the artery, allowing blood to flow. A stent is often placed at the site of blockage to permanently open the artery.
  Other Names: percutaneous coronary intervention

SUMMARY:
To study whether renal sympathetic denervation(RSD) will reduce the all-cause mortality and the recurrence rate of a composite of cardiovascular event(including angina, myocardial infarction, repeat percutaneous coronary intervention and coronary artery bypass grafting) in patients after percutaneous coronary intervention(PCI). Besides whether RSD can reduce the risk factors for coronary heart disease.

DETAILED DESCRIPTION:
Coronary heart disease is the leading cause of death worldwide, contributing to over 7.2 million deaths annually. The main measures of secondary prevention of coronary heart disease are optimizing drug therapy and changing lifestyle. optimizing drug therapy, including aspirin, beta receptor blockers, lipid regulating drugs (mostly statins, a small part fibrates) and vascular angiotensin-converting enzyme inhibitors. However, the situation for secondary prevention of coronary heart disease is not satisfying. EuroASPIRE III survey found that despite effective drug used in the primary or secondary prevention of coronary heart disease, coronary heart disease risk factors, such as high blood glucose,hypertension, high cholesterol and obesity, are still poorly controlled. At the same time sympathetic activation plays an extremely important role in the development of coronary heart disease, and high sympathetic activity after acute myocardial infarction is closely related to malignant arrhythmia and heart failure. Recently, many clinical researches have verified that catheter-based renal sympathetic denervation(RSD) can safely be used to substantially reduce blood pressure, reduce left ventricular hypertrophy, improve glucose tolerance and sleep apnea severity. Simultaneously, a marked reduction in muscle and whole-body sympathetic-nerve activity(MSNA) is apparent, with a decrease in renal and whole-body norepinephrine spillover. Hypertension, diabetes, high norepinephrine level and obstructive sleep apnea are all recognized as risk factors for the development and recurrence of coronary heart disease. So, we design this randomized parallel control clinical study to demonstrate whether RSD can reduce the mortality and the recurrence rate of a composite of cardiovascular event in patients after PCI, besides whether RSD can reduce the risk factors for coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is ≥ 18 and ≤75 years of age.
2. Individual has a clear history of coronary heart disease,and need underwent percutaneous coronary intervention .
3. Blood pressure >115/75mmHg.
4. Individual's cardiac function is between Ⅰ~Ⅲ level(NYHA)
5. Individual agrees to have all study procedures performed, and is competent and willing to provide written, informed consent to participate in this clinical study

Exclusion Criteria:

1. Individual has hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous.
2. Individual has experienced renal artery stenosis,or A history of prior renal artery intervention including balloon angioplasty or stenting. or ineligible conditions through renal artery Computed Tomography Angiogram(CTA) inspection, such as double renal artery on one side,renal artery length≤2cm, diameter≤4mm, and distortion at incept sect.
3. Individual has an estimated glomerular filtration rate (eGFR) of < 45mL/min/1.73m2, using the MDRD calculation.
4. Individual has Acute heart failure.
5. Individual has experienced a cerebrovascular accident within 3 months of the screening visit, or has widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques.
6. Individual has experienced sick sinus syndrome.
7. Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, hemophilia, or significant anemia, or arrhythmias such as atrial fibrillation).
8. Individual is pregnant, nursing or planning to be pregnant. [Female participants of childbearing potential must have a negative serum or urine human chorionic gonadotropin (hCG) pregnancy test prior to treatment.]
9. Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
10. Individual is currently enrolled in another investigational drug or device trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 24 months
  To study the effect of renal sympathetic denervation(RSD) on all-cause mortality in patients after PCI

SECONDARY OUTCOMES:
Recurrent angina pectoris | 24 months
  Previous symptoms of myocardial ischemia in patients relapsed or aggravated during follow-up, or ECG ST segment depressed compared with preoperative, or need to increase the dose of antianginal drug.
Myocardial infarction | 24 months
  It can be diagnosed by symptoms, ECG and myocardial markers changes.
Vascular recanalization again | 24 months
  Coronary angiography shows new stenosis during the follow-up and patients need PCI or coronary artery bypass grafting(CABG) again.
Chronic heart failure | 24 months
  To study whether RSD can improve the patients' heart function. And it will be judged by the NYHA classification,BNP and echocardiography.
Arrhythmia | 24 months
  If a new arrhythmia is discovered during the follow-up,it will be recorded. Patients may have symptoms of flustered, palpitations, dizziness, amaurosis, syncope and so on, which can be diagnosed by ECG and Holter.
Stroke | 24 months
  During the follow-up if a new stroke occured,it will be recorded. And it can be diagnosed by symptoms, cranial CT or MRI.
Blood pressure | 24 months
  To study the effect of renal sympathetic denervation on blood pressure in patients with hypertension,which can be measured by ambulatory blood pressure.
Blood sugar | 24 months
  In order to study whether RSD can reduce the blood sugar level and insulin resistance of diabetic patients. It will be measured by fasting blood glucose, glycated hemoglobin and fasting insulin.
Renal function | 24 months
  To study whether RSD can improve the patients' renal function, which will be measured by urine albumin, creatinine and urea nitrogen levels.
Pulse wave velocity | 24 months
  So as to study whether RSD can improve the patients' blood vessel elasticity, a pulse wave velocity (PWV)will be carried on.
Life quality | 24 months
  Life quality on 36-item short-form(SF-36)Health Survey Questionnaire will be carried out during the follow-up to study the patients' life quality.
Medication adherence | 24 months
  To study the patients'Medication adherence,we will record the type ,the dose and use time of drugs patients used during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Qijun Shan, professor, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China